CLINICAL TRIAL: NCT00870545
Title: Reintegration: The Role of Spouse Telephone BATTLEMIND Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda O. Nichols, Ph.D., Healthcare Education Specialist/Health Services Researcher, Memphis VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT074804
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Military Spouses; Support Groups; Stress Disorders; Combat Disorders
Keywords: spouses; social support; reintegration; families; military; post deployment; OEF/OIF
MeSH Terms: conditions — Stress Disorders, Traumatic; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telephone support (Experimental): 12 telephone support group sessions based on the letters of the word BATTLEMIND
  Interventions: Behavioral: Telephone support groups

INTERVENTIONS:
Behavioral: Telephone support groups — There was one intervention. Participants were enrolled in one of 14 telephone groups (each with a trained Group Leader and 6 participants) will focus on education, training in and practice of coping skills and cognitive restructuring (identifying and re-shaping negative and destructive thoughts), and support through 12 hour-long structured sessions. The content, modeled on Soldier BATTLEMIND, targets readjustment concepts based on the letters of BATTLEMIND, including Bonds, Adding and subtracting family roles, Taking control, Talking it out, Loyalty and commitment, Emotional balance, Mental health and readiness, Independence and interdependence, Navigating the system, Denial of self and a concluding session entitled Moving forward.

SUMMARY:
This study will expand the Department of Defense (DoD) one time, face-to-face post deployment BATTLEMIND training for spouses of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Guard/Reserve service members into year-long, telephone groups focusing on education, skills building and support. The goal is to build spouses' resilience to cope with reintegration, help them serve as a support system for returning service members, and ease the transition for families post-deployment.

ELIGIBILITY:
Inclusion Criteria:

1. have a spouse who participated in OEF/OIF and is at least 1 month post-deployment;
2. if not married, must have lived as married for at least one year;
3. live with the service member when not deployed;
4. have been a spouse/significant other throughout the service member's deployment period;
5. and have a telephone.

Exclusion Criteria:

1. current diagnosis of schizophrenia or other major mental illness;
2. auditory impairment that would make telephone use difficult; or
3. service member refusal of assent for spouse to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda O Nichols, PhD, Principal Investigator — Memphis VA Medical Center
Locations (1):
- Memphis VA Medical Center, Memphis, Tennessee, United States

REFERENCES:
- See also: Information and contacts — http://www.memphis.va.gov/spousebattlemind/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 2009 - January 2010 and April 2010 - June 2010. There were 86 spouses enrolled in 14 groups. Spouses were recruited nationally through online methods such as websites and emails, mailings, and referrals from military, advocacy groups and veterans facilities. Twenty-six were referrals from the national Wounded Warrior Project office.
Groups:
- Telephone Support: There was one intervention. Participants were enrolled in one of 14 telephone groups (each with a trained Group Leader and 6 participants) will focus on education, training in and practice of coping skills and cognitive restructuring (identifying and re-shaping negative and destructive thoughts), and support through 12 hour-long structured sessions. The content, modeled on Soldier BATTLEMIND, targets readjustment concepts based on the letters of BATTLEMIND, including Bonds, Adding and subtracting family roles, Taking control, Talking it out, Loyalty and commitment, Emotional balance, Mental health and readiness, Independence and interdependence, Navigating the system, Denial of self and a concluding session entitled Moving forward.
Period: Overall Study
Arm/Group | Telephone Support
Started | 86
Completed | 69
Not Completed | 17

BASELINE CHARACTERISTICS:
Groups:
- Telephone Support: 12 telephone support groups based on the letters of the word BATTLEMIND
  Telephone support groups : 12 hour-long structured telephone groups (each with a trained Group Leader and 6 participants) will focus on education, training in and practice of coping skills and cognitive restructuring (identifying and re-shaping negative and destructive thoughts), and support. The content, modeled on Soldier BATTLEMIND, targets readjustment concepts based on the letters of BATTLEMIND.
Arm/Group | Telephone Support
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Spouse Self-report of Depression
Description: Depression measured with the Patient Health Questionnaire (PHQ)-9 at baseline, six and 12 months. Scores range from 0-27 with lower scores indicating less depressive symptoms.
Time Frame: Baseline, 6 months, and 12 months
Population: All participants with depression data at baseline, six and twelve months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 86
units on a scale
  Depression score at baseline (n=86) | 8.9 (5.9)
  Depression score at 6 months (n=77) | 7.4 (5.6)
  Depression score at 12 months (n=70) | 6.9 (5.7)
Statistical Analysis 1: Comparison: Telephone Support; Change in scores measured across three time points (baseline, 6 and 12 months); Test type: Superiority or Other; p = .003, Mixed Models Analysis — P values less than or equal to .05 were considered statistically significant, and those between .05 and .10 were considered to document trends that approached, but did not attain, statistical significance

2. Secondary Outcome: Family Coping
Description: Family problem solving measured at baseline, six and 12 months with the F-COPES measure. Scores range from 29-145 with higher scores indicating better coping.
Time Frame: Baseline, 6 months and 12 months
Population: All participants with family coping data at baseline, six and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 85
units on a scale
  Family coping score at baseline (n=85) | 104.3 (13.8)
  Family coping score at 6 months (n=77) | 104.7 (13.7)
  Family coping score at 12 months (n=70) | 105.7 (14.5)
Statistical Analysis 1: Comparison: Telephone Support; Analysis was change in score over time (baseline, 6 and 12 months); Test type: Superiority or Other; p = .20, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Anxiety
Description: Anxiety measured with the Generalized Anxiety Disorder -7 (GAD-7)measured at baseline, six and 12 months. Scores range from 0-21, with lower scores indicating fewer anxiety symptoms.
Time Frame: baseline, 6 months and 12 months
Population: All participants with anxiety scores at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 86
units on a scale
  Anxiety score at baseline (n=86) | 8.9 (5.7)
  Anxiety score at 6 months (n=77) | 6.7 (5.1)
  Anxiety score at 12 months (n=70) | 6.7 (5.6)
Statistical Analysis 1: Comparison: Telephone Support; Change in scores measured across three time points (baseline, 6 and 12 months); Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Quality of Marriage
Description: Measure of marriage quality using Quality Marriage Index at baseline, six and 12 months. Scores range from 6-45 with higher scores indicating better quality of marriage.
Time Frame: Baseline, 6 and 12 months
Population: All participants with quality marriage index scores at the three time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 86
units on a scale
  Marriage quality score at baseline (n=86) | 32.7 (8.0)
  Marriage quality score at 6 months (n=77) | 31.6 (9.9)
  Marriage quality score at 12 months (n=70) | 31.9 (9.8)
Statistical Analysis 1: Comparison: Telephone Support; Analysis was change in score over time (baseline, 6 months, 12 months); Test type: Superiority or Other; p = .26, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Spouse Social Support
Description: Support measured with the Social Support Index at baseline, six and 12 months. Scores range from 0-68 with higher scores indicating better social support.
Time Frame: baseline, 6 months, and 12 months
Population: All participants with social support data at baseline, six and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 86
units on a scale
  Social Support score at baseline (n=86) | 44.0 (8.6)
  Social Support score at 6 months (n=77) | 46.0 (10.2)
  Social Support score at 12 months (n=70) | 45.5 (10.1)
Statistical Analysis 1: Comparison: Telephone Support; Analysis was change in scores over time (baseline, 6 months, and 12 months); Test type: Superiority or Other; p = .04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Family Communication
Description: Family communication measured with the Family Problem Solving Communication scale at baseline, six and 12 months. Scores range from 0-30 with higher scores indicating better communication.
Time Frame: baseline, 6 months, and 12 months
Population: All participants with family communication data at baseline, six and 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone Support
Number analyzed (Participants) | 85
units on a scale
  Family communication score at baseline (n=85) | 19.9 (6.2)
  Family communication score at 6 months (n=77) | 20.9 (6.4)
  Family communication score at 12 months (n=70) | 20.9 (6.2)
Statistical Analysis 1: Comparison: Telephone Support; Analysis was change in score over time (baseline, 6 months, and 12 months); Test type: Superiority or Other; p = .10, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Telephone Support
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

LIMITATIONS AND CAVEATS:
Small sample size, some of the Wounded Warrior Project spouses knew each other, pilot feasibility study and not a randomized controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No